CLINICAL TRIAL: NCT04133038
Title: Assessment of Feeding and Eating Disorders of Young Children : Standardisation of a New Tool, the Hetero-questionnaire Named ORALQUEST
Brief Title: Evaluation of ORALQUEST
Acronym: ORALQUEST
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Filiere de Sante Maladies Rares TETECOU (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190790; 2019-A01215-52 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-10-18; First posted 2019-10-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Feeding and Eating Disorders of Childhood
Keywords: Feeding disorders; Eating disorders; Evaluation
MeSH Terms: conditions — Feeding and Eating Disorders of Childhood; Feeding and Eating Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Children consulting: Children consulting in the expert center for food difficulties.
  Interventions: Other: Questionnaire
- Pierre Robin sequence: Children with Pierre Robin sequence following for food difficulties.
  Interventions: Other: Questionnaire
- Cardiac malformations: Children with cardiac malformations followed for food difficulties.
  Interventions: Other: Questionnaire
- Oesophageal atresia: Children with oesophageal atresia followed for food difficulties.
  Interventions: Other: Questionnaire
- Cleft lip and palate: Children with cleft lip and palate followed for food difficulties.
  Interventions: Other: Questionnaire
- Autism spectrum disorders: Children followed for congenital pathology that cause food difficulties.
  Interventions: Other: Questionnaire
- Ex-prematurity < 32 AG: Children born premature followed for food difficulties.
  Interventions: Other: Questionnaire
- Chromosomal anomalies: Children with chromosomal anomalies followed for food difficulties.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Parent(s) answering questionnaires about his child's phobic and selective eating behaviour.

SUMMARY:
Feeding and eating disorders are frequent in children of the general population. They are much more frequent in children with congenital chronic diseases. The analysis of feeding and eating disorders in children is difficult since their causes are complex and multiple. In addition to the clinical examination and the instrumental investigation, a parental questionnaire is very useful in assessing these disorders. The questionnaire (testing the right period of age, evaluating the 4 aspects involved in the disorders, translated in French) does not exist. Consequently, the Necker team of the reference center, has built a hetero-questionnaire named ORALQUEST, which analyses 4 dimensions of the feeding and eating disorders of young children from 9 months to 6 years: behaviour, oral motor skills, sensory sensitivity and familial environment.

The objective of the study is to test the metrological qualities of Oralquest in children with congenital chronic diseases including feeding and eating disorders.

The questionnaire will be proposed to 7 cohorts of children who are followed in Necker for :

* oesophageal atresia,
* cardiac malformations,
* Pierre Robin sequence,
* cleft lip and palate,
* autism spectrum disorders,
* ex-prematurity < 32 AG,
* chromosomal anomalies, and proposed to children consulting in the expert center for phobic and selective eating behaviour.

The analysis of the metrological qualities of the questionnaire include several calculation and specialized methods: inter-rate concordance; test-retest; intrinsic validity, concurrent validity, sensitivity/specificity.

DETAILED DESCRIPTION:
Objectives of the study To analyse the properties of a new scale that evaluates feeding and eating disorders of young children. This scale is a hetero-questionnaire that was build by an expert team. It includes 46 questions scored with a Likert scale. These questions identify 4 fields: behaviour during the meal, oromotor skills, sensory sensitivity and familial environment. Each field gives a sub-score, their addition gives a global score

Methods

To evaluate the metrological qualities of this questionnaire, the investigators are going to investigate 300 children followed-up in Necker for either Aversive/restrictive food intake disorders (ARFID) or for chronic congenital disease very often complicated with feeding and eating disorders:

* oesophageal atresia,
* cardiac malformations,
* Pierre Robin sequence,
* cleft lip and palate,
* autism spectrum disorders,
* ex-prematurity < 32 AG,
* chromosomal anomalies,

They want to test the statistical significance of the score. For that, they will test:

* the face validity,
* the structure validity
* and, the internal consistence of Oralquest. The interconcept validity will be analysed by comparing the Oralquest results to the best gold standard tests that are found for each field tested by Oralquest.

For the global score : The screening test : self-questionnaire, the Montreal Children Feeding Scale.

For the behavior score : the symptom check list (items regarding eating). For the oromotor skills : (Schedule for Oral-Motor Assessment) for the children aged 9-24 months and the Oral-Motor Assessment Scale for the children aged 2-6 years).

For the familial environment : The STAI (State Trait Anxiety Inventory).

The reproductibility will be tested by :

* Test-retest
* Inter examiner reproductibility
* sensibility
* specificity

ELIGIBILITY:
Inclusion Criteria:

- child of 9 months to 6 years old:

* Consulting for food difficulties in the expert center for phobic and selective eating behaviour of Necker-Enfants malades hospital or
* Followed to Necker-Enfants Malades hospital for one of 7 chronic congenital pathologies: oesophageal atresia, cardiac malformations, Pierre Robin sequence, cleft lip and palate, autism spectrum disorders, ex-prematurity < 32 AG, chromosomal anomalies

Exclusion Criteria:

- parent (s) with a low level of French to understand the questions

Ages: 9 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 9 months to 6 years with or without a congenital disease with a phobic and selective eating behaviour.
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Validity of ORALQUEST questionnaire | 1 month
  Metrological qualities including the face validity, the structure validity and, the internal consistency and the interconcept validity of ORALQUEST.

SECONDARY OUTCOMES:
ORALQUEST global score | 1 day
  ORALQUEST global score in each of the 8 cohorts of children
Behaviour during the meal ORALQUEST Sub-score | 1 day
  ORALQUEST sub-score in each of the 8 cohorts of children
Oromotor skills ORALQUEST Sub-score | 1 day
  ORALQUEST sub-score in each of the 8 cohorts of children
Sensory sensitivity ORALQUEST Sub-score | 1 day
  ORALQUEST sub-score in each of the 8 cohorts of children
Familial environment ORALQUEST Sub-score | 1 day
  ORALQUEST sub-score in each of the 8 cohorts of children

CONTACTS AND LOCATIONS:
Overall Officials: Véronique ABADIE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Pediatry, Necker-Enfants Malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No